CLINICAL TRIAL: NCT03049488
Title: VRC 317: A Phase I Randomized, Open-Label Clinical Trial to Evaluate Dose, Safety, Tolerability and Immunogenicity of a Stabilized Prefusion RSV F Subunit Protein Vaccine, VRC-RSVRGP084-00-VP (DS-Cav1), Alone or With Alum Adjuvant, in Healthy Adults
Brief Title: Dose, Safety, Tolerability and Immunogenicity of a Stabilized Prefusion RSV F Subunit Protein Vaccine, VRC-RSVRGP084-00-VP (DS-Cav1), Alone or With Alum Adjuvant, in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 170058; 17-I-0058 (Other: NIH NIAID IRB)
Record Dates: First submitted 2017-02-09; First posted 2017-02-10 (Actual); Results first posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Respiratory Syncytial Virus
Keywords: Immune Response; Respiratory Syncytial Virus; Vaccine-Mediated Protection; Neutralizing Antibody; Antibody Response
MeSH Terms: interventions — aluminum sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1: DS-Cav1 (50 mcg) (Experimental): DS-Cav1 (50 mcg) administered intramuscularly (IM) by Needle/Syringe (Day 0 and Week 12*)
  *To evaluate the safety or immunogenicity of a single vaccine dose, the Week 12 dose was optional for the last 5 subjects who enrolled in this group and received the Day 0 injection.
  Interventions: Biological: VRC-RSVRGP084-00-VP
- Group 2: DS-Cav1 (50 mcg) + alum (Experimental): DS-Cav1 (50 mcg) + alum administered IM by Needle/Syringe (Day 0 and Week 12*)
  *To evaluate the safety or immunogenicity of a single vaccine dose, the Week 12 dose was optional for the last 5 subjects who enrolled in this group and received the Day 0 injection.
  Interventions: Biological: VRC-RSVRGP084-00-VP; Other: Aluminum Hydroxide Suspension
- Group 3: DS-Cav1 (150 mcg) (Experimental): DS-Cav1 (150 mcg) administered IM by Needle/Syringe (Day 0 and Week 12*)
  *The Week 12 dose was optional for the last 5 subjects who enrolled in this group and received the Day 0 injection, and for 5 additional subjects who were enrolled to evaluate the safety or immunogenicity of a single vaccine dose.
  Interventions: Biological: VRC-RSVRGP084-00-VP
- Group 4: DS-Cav1 (150 mcg) + alum (Experimental): DS-Cav1 (150 mcg) + alum administered IM by Needle/Syringe (Day 0 and Week 12*)
  *To evaluate the safety or immunogenicity of a single vaccine dose, the Week 12 dose was optional for the last 5 subjects who enrolled in this group and received the Day 0 injection.
  Interventions: Biological: VRC-RSVRGP084-00-VP; Other: Aluminum Hydroxide Suspension
- Group 5: DS-Cav1 (500 mcg) (Experimental): DS-Cav1 (500 mcg) administered IM by Needle/Syringe (Day 0 and Week 12*)
  *To evaluate the safety or immunogenicity of a single vaccine dose, the Week 12 dose was optional for the last 5 subjects who enrolled in this group and received the Day 0 injection.
  Interventions: Biological: VRC-RSVRGP084-00-VP
- Group 6:DS-Cav1 (500 mcg) + alum (Experimental): DS-Cav1 (500 mcg) + alum administered IM by Needle/Syringe (Day 0 and Week 12*)
  *To evaluate the safety or immunogenicity of a single vaccine dose, the Week 12 dose was optional for the last 5 subjects who enrolled in this group and received the Day 0 injection.
  Interventions: Biological: VRC-RSVRGP084-00-VP; Other: Aluminum Hydroxide Suspension

INTERVENTIONS:
Biological: VRC-RSVRGP084-00-VP — VRC-RSVRGP084-00-VP is an investigational respiratory syncytial virus (RSV) vaccine.
  Other Names: DS-Cav1
Other: Aluminum Hydroxide Suspension — Aluminum Hydroxide Suspension, alum, is an adjuvant.
  Other Names: Alum
  Arms: Group 2: DS-Cav1 (50 mcg) + alum; Group 4: DS-Cav1 (150 mcg) + alum; Group 6:DS-Cav1 (500 mcg) + alum

SUMMARY:
Background:

Respiratory Syncytial Virus (RSV) is a virus that infects the lungs and breathing passages. Healthy adults who are infected generally have mild cold symptoms for a week or two. But it can also be serious, especially for infants and older adults. It can be spread by direct or indirect contact with respiratory secretions. Researchers want to study a new vaccine to prevent RSV.

Objective:

To see if a vaccine for RSV is safe and if it causes side effects.

Eligibility:

Healthy adults 18-50 years old

Design:

Volunteers were screened in a separate screening protocol.

Subjects had 13 visits over 1 year.

Some subjects received just vaccine. Some received vaccine mixed with alum adjuvant.

All subjects received their dose by injection in the upper arm. They received up to two doses, one at the beginning of the study and another 12 weeks later.

Subjects were monitored for 1 hour after injection and called to check on their safety 1 day after.

Subjects recorded their temperature and side effects for 7 days after each vaccination.

Subjects were provided with a thermometer to measure their temperature and a ruler to measure any changes if these occurred on their skin at the injection site.

At all visits, subjects were checked for health changes or problems. They may have had blood drawn.

At some visits, subjects had samples collected from their nose and mouth.

DETAILED DESCRIPTION:
Study Design:

This is a Phase I, open-label, dose escalation study to evaluate the dose, safety, tolerability, and immunogenicity of VRC-RSVRGP084-00-VP vaccine alone or with alum adjuvant in a 2-injection regimen. The hypotheses are that the vaccine will be safe and tolerable for human administration, and will induce detectable immune response. The primary objective is to evaluate the safety and tolerability of the investigational vaccine at 3 dose levels administered alone or with alum adjuvant in healthy adults. Secondary objectives relate to humoral and cellular immunogenicity of the investigational vaccine regimen.

Product Description:

VRC-RSVRGP084-00-VP (DS-Cav1) was developed by VRC, NIAID and is composed of the respiratory syncytial virus (RSV) fusion (F) glycoprotein ectodomain assembled as a trimer stabilized in its prefusion native conformation with a foldon trimerization domain at the C-terminus and 4 internal mutations designated DS-Cav1 (4.1DHFR_RSVAF). The sequence is based on the RSV A2 strain from subtype A. The product was provided at a concentration of 0.5 mg/mL in 3 mL glass vials filled to 1.2 mL. Adjuvant was an aluminum hydroxide suspension (alum) provided in a sterile, pyrogen-free suspension at a concentration of 5 mg/mL in 3 mL glass vials filled to 0.7 mL. The alum dose was 500 mcg and was field mixed.

Subjects:

Healthy adult subjects ages 18-50 years

Study Plan:

Subjects were randomized into DS-Cav1 or DS-Cav1 plus alum in each dose during the study. Dose continuation and dose escalation evaluations occurred to ensure the safety data support proceeding to the higher doses. Subjects were evaluated for safety and immune responses through blood and mucosal sample collection at specified timepoints throughout the study.

VRC 317 Study Schema:

* Group: 1; Subjects: 15; Dose: 50mcg; Day 0: DS-Cav1; Week 12 [1]: DS-Cav1
* Group: 2; Subjects: 15; Dose: 50mcg; Day 0: DS-Cav1 + alum; Week 12 [1]: DS-Cav1 + alum
* Group: 3; Subjects: 15; Dose: 150mcg; Day 0: DS-Cav1; Week 12 [1]: DS-Cav1
* Group: 4; Subjects: 15; Dose: 150mcg; Day 0: DS-Cav1 + alum; Week 12 [1]: DS-Cav1 + alum
* Group: 5; Subjects: 15; Dose: 500mcg; Day 0: DS-Cav;1 Week 12 [1]: DS-Cav1
* Group: 6; Subjects: 15; Dose: 500mcg; Day 0: DS-Cav1 + alum; Week 12 [1]: DS-Cav1 + alum

All DS-Cav1 vaccinations were administered with needle and syringe into the deltoid muscle.

Total Planned Subjects: 90 (Up to 100 subjects could have been enrolled if needed to evaluate safety or immunogenicity.)

• [1] Week 12 dose: Optional for the last 5 subjects enrolled in each group who received the Day 0 injection and any additional subjects needed to evaluate safety or immunogenicity of a single injection.

Duration:

The study schedule required 13 clinic visits and a telephone contact after each injection.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. 18 to 50 years of age.
  2. Willing and able to complete the informed consent process.
  3. Available for clinic visits through 44 weeks after enrollment.
  4. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
  5. Willing to donate blood and mucosal samples to be stored and used for future research.
  6. In good general health without clinically significant medical history.
  7. Physical examination and laboratory results without clinically significant findings and a Body Mass Index (BMI) less than or equal to 40 within the 56 days prior to enrollment. Laboratory criteria within 56 days prior to enrollment:
  8. White Blood Cell (WBC) and differential either within institutional normal range or accompanied by Principal Investigator (PI) or designee approval.
  9. Platelets = 125,000-500,000/mm^3.
  10. Hemoglobin within institutional normal range.
  11. Creatinine less than or equal to 1.1 x upper limit of normal (ULN).
  12. Alanine aminotransferase (ALT) less than or equal to 1.25 x ULN.
  13. Negative for HIV infection by an FDA approved method of detection.

      Criteria applicable to women of childbearing potential:
  14. Negative result on a human chorionic gonadotropin pregnancy test on day of enrollment before receiving study product.
  15. Agree to use effective means of birth control from at least 21 days before enrollment through 4 weeks after the last injection.
* EXCLUSION CRITERIA:

Criteria applicable to women of childbearing potential:

1. Breast-feeding or planning to become pregnant through 4 weeks after the last injection.

   Subject has received any of the following:
2. More than 10 days of systemic immunosuppressive medications or cytotoxic medications within the 4 weeks prior to enrollment or any within the 14 days prior to enrollment.
3. Blood products within 16 weeks prior to enrollment.
4. Live attenuated vaccines within 4 weeks prior to enrollment.
5. Inactivated vaccines within 2 weeks prior to enrollment.
6. Investigational research agents within 4 weeks prior to enrollment or planning to receive investigational products while on the study.
7. Current allergen immunotherapy with antigen injections, unless on maintenance schedule.
8. Current anti-tuberculosis(TB) prophylaxis or therapy.

   Subject has any of the following:
9. Serious reactions to vaccines that preclude receipt of study injections as determined by the investigator.
10. Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema.
11. Asthma that is not well controlled.
12. Diabetes mellitus (type I or II), with the exception of gestational diabetes.
13. Thyroid disease that is not well controlled.
14. Hypertension that is not well controlled.
15. Evidence of autoimmune disease or immunodeficiency.
16. Idiopathic urticaria within the past year.
17. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
18. Malignancy that is active or history of malignancy that is likely to recur during the study.
19. Seizure disorder other than: 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the last 3 years.
20. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.
21. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; or within 5 years prior to enrollment, a history of suicide plan or attempt.
22. Any medical, psychiatric, or social condition that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a subject s ability to give informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace L Chen, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruckwardt TJ, Morabito KM, Graham BS. Determinants of early life immune responses to RSV infection. Curr Opin Virol. 2016 Feb;16:151-157. doi: 10.1016/j.coviro.2016.01.003. Epub 2016 Mar 15. PMID 26986236
- [Background] Ngwuta JO, Chen M, Modjarrad K, Joyce MG, Kanekiyo M, Kumar A, Yassine HM, Moin SM, Killikelly AM, Chuang GY, Druz A, Georgiev IS, Rundlet EJ, Sastry M, Stewart-Jones GB, Yang Y, Zhang B, Nason MC, Capella C, Peeples ME, Ledgerwood JE, McLellan JS, Kwong PD, Graham BS. Prefusion F-specific antibodies determine the magnitude of RSV neutralizing activity in human sera. Sci Transl Med. 2015 Oct 14;7(309):309ra162. doi: 10.1126/scitranslmed.aac4241. PMID 26468324
- [Background] Graham BS, Modjarrad K, McLellan JS. Novel antigens for RSV vaccines. Curr Opin Immunol. 2015 Aug;35:30-8. doi: 10.1016/j.coi.2015.04.005. Epub 2015 Jun 10. PMID 26070108
- [Background] Crank MC, Ruckwardt TJ, Chen M, Morabito KM, Phung E, Costner PJ, Holman LA, Hickman SP, Berkowitz NM, Gordon IJ, Yamshchikov GV, Gaudinski MR, Kumar A, Chang LA, Moin SM, Hill JP, DiPiazza AT, Schwartz RM, Kueltzo L, Cooper JW, Chen P, Stein JA, Carlton K, Gall JG, Nason MC, Kwong PD, Chen GL, Mascola JR, McLellan JS, Ledgerwood JE, Graham BS; VRC 317 Study Team. A proof of concept for structure-based vaccine design targeting RSV in humans. Science. 2019 Aug 2;365(6452):505-509. doi: 10.1126/science.aav9033. PMID 31371616
- [Derived] Chang LA, Phung E, Crank MC, Morabito KM, Villafana T, Dubovsky F, Falloon J, Esser MT, Lin BC, Chen GL, Graham BS, Ruckwardt TJ. A prefusion-stabilized RSV F subunit vaccine elicits B cell responses with greater breadth and potency than a postfusion F vaccine. Sci Transl Med. 2022 Dec 21;14(676):eade0424. doi: 10.1126/scitranslmed.ade0424. Epub 2022 Dec 21. PMID 36542692
- [Derived] Ruckwardt TJ, Morabito KM, Phung E, Crank MC, Costner PJ, Holman LA, Chang LA, Hickman SP, Berkowitz NM, Gordon IJ, Yamshchikov GV, Gaudinski MR, Lin B, Bailer R, Chen M, Ortega-Villa AM, Nguyen T, Kumar A, Schwartz RM, Kueltzo LA, Stein JA, Carlton K, Gall JG, Nason MC, Mascola JR, Chen G, Graham BS; VRC 317 study team. Safety, tolerability, and immunogenicity of the respiratory syncytial virus prefusion F subunit vaccine DS-Cav1: a phase 1, randomised, open-label, dose-escalation clinical trial. Lancet Respir Med. 2021 Oct;9(10):1111-1120. doi: 10.1016/S2213-2600(21)00098-9. Epub 2021 Apr 14. PMID 33864736
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-I-0058.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults were recruited from the Washington, D.C., metropolitan area.
Groups:
- Group 1: DS-Cav1 (50 mcg): DS-Cav1 (50 mcg) administered intramuscularly (IM) by Needle/Syringe (Day 0 and Week 12*)
  *To evaluate the safety or immunogenicity of a single vaccine dose, the Week 12 dose was optional for the last 5 subjects who enrolled in this group and received the Day 0 injection.
  VRC-RSVRGP084-00-VP: VRC-RSVRGP084-00-VP is an investigational respiratory syncytial virus (RSV) vaccine.
- Group 2: DS-Cav1 (50 mcg) + Alum: DS-Cav1 (50 mcg) + alum administered IM by Needle/Syringe (Day 0 and Week 12*)
  *To evaluate the safety or immunogenicity of a single vaccine dose, the Week 12 dose was optional for the last 5 subjects who enrolled in this group and received the Day 0 injection.
  VRC-RSVRGP084-00-VP: VRC-RSVRGP084-00-VP is an investigational respiratory syncytial virus (RSV) vaccine.
  Aluminum Hydroxide Suspension: Aluminum Hydroxide Suspension, alum, is an adjuvant.
- Group 3: DS-Cav1 (150 mcg): DS-Cav1 (150 mcg) administered IM by Needle/Syringe (Day 0 and Week 12*)
  *The Week 12 dose was optional for the last 5 subjects who enrolled in this group and received the Day 0 injection, and for 5 additional subjects who were enrolled to evaluate the safety or immunogenicity of a single vaccine dose.
  VRC-RSVRGP084-00-VP: VRC-RSVRGP084-00-VP is an investigational respiratory syncytial virus (RSV) vaccine.
- Group 4: DS-Cav1 (150 mcg) + Alum: DS-Cav1 (150 mcg) + alum administered IM by Needle/Syringe (Day 0 and Week 12*)
  *To evaluate the safety or immunogenicity of a single vaccine dose, the Week 12 dose was optional for the last 5 subjects who enrolled in this group and received the Day 0 injection.
  VRC-RSVRGP084-00-VP: VRC-RSVRGP084-00-VP is an investigational respiratory syncytial virus (RSV) vaccine.
  Aluminum Hydroxide Suspension: Aluminum Hydroxide Suspension, alum, is an adjuvant.
- Group 5: DS-Cav1 (500 mcg): DS-Cav1 (500 mcg) administered IM by Needle/Syringe (Day 0 and Week 12*)
  *To evaluate the safety or immunogenicity of a single vaccine dose, the Week 12 dose was optional for the last 5 subjects who enrolled in this group and received the Day 0 injection.
  VRC-RSVRGP084-00-VP: VRC-RSVRGP084-00-VP is an investigational respiratory syncytial virus (RSV) vaccine.
- Group 6: DS-Cav1 (500 mcg) + Alum: DS-Cav1 (500 mcg) + alum administered IM by Needle/Syringe (Day 0 and Week 12*)
  *To evaluate the safety or immunogenicity of a single vaccine dose, the Week 12 dose was optional for the last 5 subjects who enrolled in this group and received the Day 0 injection.
  VRC-RSVRGP084-00-VP: VRC-RSVRGP084-00-VP is an investigational respiratory syncytial virus (RSV) vaccine.
  Aluminum Hydroxide Suspension: Aluminum Hydroxide Suspension, alum, is an adjuvant.
Period: Overall Study
Arm/Group | Group 1: DS-Cav1 (50 mcg) | Group 2: DS-Cav1 (50 mcg) + Alum | Group 3: DS-Cav1 (150 mcg) | Group 4: DS-Cav1 (150 mcg) + Alum | Group 5: DS-Cav1 (500 mcg) | Group 6: DS-Cav1 (500 mcg) + Alum
Started | 15 | 15 | 20 | 15 | 15 | 15
Received First Product Administration | 15 | 15 | 20 | 15 | 15 | 15
Received Optional Second Dose | 10 | 11 | 11 | 9 | 11 | 10
Completed | 13 | 13 | 20 | 13 | 13 | 15
Not Completed | 2 | 2 | 0 | 2 | 2 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Moved from Area | 1 | 0 | 0 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Population includes all enrolled subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: DS-Cav1 (50 mcg) | Group 2: DS-Cav1 (50 mcg) + Alum | Group 3: DS-Cav1 (150 mcg) | Group 4: DS-Cav1 (150 mcg) + Alum | Group 5: DS-Cav1 (500 mcg) | Group 6: DS-Cav1 (500 mcg) + Alum | Total
Number analyzed (Participants) | 15 | 15 | 20 | 15 | 15 | 15 | 95
Age, Customized [Count of Participants; unit: Participants]
  18-20 years | 0 | 2 | 1 | 1 | 0 | 0 | 4
  21-30 years | 4 | 4 | 9 | 6 | 8 | 11 | 42
  31-40 years | 9 | 5 | 6 | 6 | 4 | 3 | 33
  41-50 years | 2 | 4 | 4 | 2 | 3 | 1 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 9 | 8 | 9 | 8 | 49
  Male | 6 | 9 | 11 | 7 | 6 | 7 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 1 | 4 | 0 | 3 | 3 | 15
  Black or African American | 1 | 3 | 1 | 4 | 0 | 0 | 9
  White | 10 | 11 | 13 | 9 | 12 | 10 | 65
  Multiracial | 0 | 0 | 2 | 2 | 0 | 2 | 6
  Hispanic/Latino | 0 | 1 | 2 | 0 | 4 | 1 | 8
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  18.5-24.9 kg/m^2 | 5 | 6 | 8 | 5 | 7 | 8 | 39
  25.0-29.9 kg/m^2 | 8 | 3 | 9 | 7 | 7 | 5 | 39
  30.0 kg/m^2 or over | 2 | 6 | 3 | 3 | 1 | 2 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Local Reactogenicity Signs and Symptoms Within 7 Days of the First Product Administration of DS-Cav1 Alone or With Alum Adjuvant
Description: Subjects recorded the occurrence of solicited symptoms on a diary card for 7 days after the first study product administration and reviewed the diary card with clinic staff at a follow up visit. Subjects were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of subjects reporting any local symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA Guidance - September 2007).
Time Frame: 7 days after the first product administration (Day 7)
Population: Population included all enrolled subjects who received at least one study injection of DS-Cav1 alone or with alum adjuvant and provided safety data (via diary card and/or laboratory results) following the injection (N=95).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DS-Cav1 (50 mcg) | Group 2: DS-Cav1 (50 mcg) + Alum | Group 3: DS-Cav1 (150 mcg) | Group 4: DS-Cav1 (150 mcg) + Alum | Group 5: DS-Cav1 (500 mcg) | Group 6: DS-Cav1 (500 mcg) + Alum
Number analyzed (Participants) | 15 | 15 | 20 | 15 | 15 | 15
Participants
  Pain/Tenderness: None | 6 | 5 | 11 | 8 | 7 | 6
  Pain/Tenderness: Mild | 9 | 10 | 9 | 7 | 8 | 9
  Pain/Tenderness: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: None | 15 | 15 | 20 | 15 | 15 | 14
  Swelling: Mild | 0 | 0 | 0 | 0 | 0 | 1
  Swelling: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Redness: None | 15 | 15 | 20 | 15 | 15 | 15
  Redness: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Redness: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Redness: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Any Local Symptom: None | 6 | 5 | 11 | 8 | 7 | 6
  Any Local Symptom: Mild | 9 | 10 | 9 | 7 | 8 | 9
  Any Local Symptom: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Any Local Symptom: Severe | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Subjects Reporting Local Reactogenicity Signs and Symptoms Within 7 Days of the Second Product Administration of DS-Cav1 Alone or With Alum Adjuvant
Description: Subjects recorded the occurrence of solicited symptoms on a diary card for 7 days after the second study product administration and reviewed the diary card with clinic staff at a follow up visit. Subjects were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of subjects reporting any local symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA Guidance - September 2007).
Time Frame: 7 days after the second product administration (Day 91)
Population: Population included all enrolled subjects who received the optional second study injection of DS-Cav1 alone or with alum adjuvant and provided safety data (via diary card and/or laboratory results) following the injection (N=62).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DS-Cav1 (50 mcg) | Group 2: DS-Cav1 (50 mcg) + Alum | Group 3: DS-Cav1 (150 mcg) | Group 4: DS-Cav1 (150 mcg) + Alum | Group 5: DS-Cav1 (500 mcg) | Group 6: DS-Cav1 (500 mcg) + Alum
Number analyzed (Participants) | 10 | 11 | 11 | 9 | 11 | 10
Participants
  Pain/Tenderness: None | 3 | 6 | 6 | 4 | 2 | 3
  Pain/Tenderness: Mild | 7 | 5 | 5 | 5 | 8 | 7
  Pain/Tenderness: Moderate | 0 | 0 | 0 | 0 | 1 | 0
  Pain/Tenderness: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: None | 10 | 11 | 11 | 9 | 11 | 10
  Swelling: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Redness: None | 10 | 11 | 11 | 9 | 11 | 10
  Redness: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Redness: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Redness: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Any Local Symptom: None | 3 | 6 | 6 | 4 | 2 | 3
  Any Local Symptom: Mild | 7 | 5 | 5 | 5 | 8 | 7
  Any Local Symptom: Moderate | 0 | 0 | 0 | 0 | 1 | 0
  Any Local Symptom: Severe | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Subjects Reporting Local Reactogenicity Signs and Symptoms Within 7 Days of Any Product Administration of DS-Cav1 Alone or With Alum Adjuvant
Description: Subjects recorded the occurrence of solicited symptoms on a diary card for 7 days after each study product administration and reviewed the diary card with clinic staff at a follow up visit. Subjects were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of subjects reporting any local symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA Guidance - September 2007).
Time Frame: 7 days after each product administration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- All DS-Cav1 Dose Groups: DS-Cav1 dose groups included adults who received up to two doses of either DS-Cav1 (50 mcg) alone, DS-Cav1 (50 mcg) + alum, DS-Cav1 (150 mcg) alone, DS-Cav1 (150 mcg) + alum, DS-Cav1 (500 mcg) alone, or DS-Cav1 (500 mcg) + alum 12 weeks apart.
Arm/Group | Group 1: DS-Cav1 (50 mcg) | Group 2: DS-Cav1 (50 mcg) + Alum | Group 3: DS-Cav1 (150 mcg) | Group 4: DS-Cav1 (150 mcg) + Alum | Group 5: DS-Cav1 (500 mcg) | Group 6: DS-Cav1 (500 mcg) + Alum | All DS-Cav1 Dose Groups
Number analyzed (Participants) | 15 | 15 | 20 | 15 | 15 | 15 | 95
Participants
  Pain/Tenderness: None | 4 | 5 | 8 | 3 | 4 | 3 | 27
  Pain/Tenderness: Mild | 11 | 10 | 12 | 12 | 10 | 12 | 67
  Pain/Tenderness: Moderate | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Pain/Tenderness: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: None | 15 | 15 | 20 | 15 | 15 | 14 | 94
  Swelling: Mild | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Swelling: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Swelling: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness: None | 15 | 15 | 20 | 15 | 15 | 15 | 95
  Redness: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Redness: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Local Symptom: None | 4 | 5 | 8 | 3 | 4 | 3 | 27
  Any Local Symptom: Mild | 11 | 10 | 12 | 12 | 10 | 12 | 67
  Any Local Symptom: Moderate | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Any Local Symptom: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Subjects Reporting Systemic Reactogenicity Signs and Symptoms Within 7 Days of the First Product Administration of DS-Cav1 Alone or With Alum Adjuvant
Description: Subjects recorded the occurrence of solicited symptoms on a diary card for 7 days after the first study product administration and reviewed the diary card with clinic staff at a follow up visit. Subjects were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of subjects reporting any systemic symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA Guidance - September 2007).
Time Frame: 7 days after the first product administration (Day 7)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DS-Cav1 (50 mcg) | Group 2: DS-Cav1 (50 mcg) + Alum | Group 3: DS-Cav1 (150 mcg) | Group 4: DS-Cav1 (150 mcg) + Alum | Group 5: DS-Cav1 (500 mcg) | Group 6: DS-Cav1 (500 mcg) + Alum
Number analyzed (Participants) | 15 | 15 | 20 | 15 | 15 | 15
Participants
  Malaise: None | 13 | 13 | 17 | 12 | 11 | 11
  Malaise: Mild | 2 | 2 | 3 | 3 | 4 | 4
  Malaise: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Malaise: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 15 | 13 | 19 | 9 | 12 | 13
  Myalgia: Mild | 0 | 2 | 1 | 6 | 3 | 2
  Myalgia: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 13 | 11 | 18 | 10 | 13 | 10
  Headache: Mild | 2 | 4 | 2 | 5 | 2 | 5
  Headache: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Headache: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 14 | 15 | 20 | 14 | 13 | 13
  Chills: Mild | 1 | 0 | 0 | 1 | 2 | 2
  Chills: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 14 | 14 | 19 | 15 | 14 | 14
  Nausea: Mild | 1 | 1 | 1 | 0 | 1 | 1
  Nausea: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: None | 15 | 15 | 20 | 15 | 14 | 15
  Temperature: Mild | 0 | 0 | 0 | 0 | 1 | 0
  Temperature: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Any Systemic Symptom: None | 12 | 11 | 15 | 9 | 10 | 9
  Any Systemic Symptom: Mild | 3 | 4 | 5 | 6 | 5 | 6
  Any Systemic Symptom: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Any Systemic Symptom: Severe | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Subjects Reporting Systemic Reactogenicity Signs and Symptoms Within 7 Days of the Second Product Administration of DS-Cav1 Alone or With Alum Adjuvant
Description: Subjects recorded the occurrence of solicited symptoms on a diary card for 7 days after the second study product administration and reviewed the diary card with clinic staff at a follow up visit. Subjects were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of subjects reporting any systemic symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA Guidance - September 2007).
Time Frame: 7 days after the second product administration (Day 91)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DS-Cav1 (50 mcg) | Group 2: DS-Cav1 (50 mcg) + Alum | Group 3: DS-Cav1 (150 mcg) | Group 4: DS-Cav1 (150 mcg) + Alum | Group 5: DS-Cav1 (500 mcg) | Group 6: DS-Cav1 (500 mcg) + Alum
Number analyzed (Participants) | 10 | 11 | 11 | 9 | 11 | 10
Participants
  Malaise: None | 9 | 9 | 11 | 8 | 8 | 9
  Malaise: Mild | 0 | 2 | 0 | 1 | 3 | 1
  Malaise: Moderate | 1 | 0 | 0 | 0 | 0 | 0
  Malaise: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 9 | 10 | 9 | 8 | 10 | 7
  Myalgia: Mild | 1 | 1 | 2 | 1 | 1 | 3
  Myalgia: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 8 | 10 | 10 | 8 | 8 | 9
  Headache: Mild | 2 | 1 | 1 | 1 | 2 | 1
  Headache: Moderate | 0 | 0 | 0 | 0 | 1 | 0
  Headache: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 10 | 11 | 11 | 9 | 11 | 9
  Chills: Mild | 0 | 0 | 0 | 0 | 0 | 1
  Chills: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 10 | 11 | 11 | 9 | 11 | 9
  Nausea: Mild | 0 | 0 | 0 | 0 | 0 | 1
  Nausea: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: None | 10 | 11 | 11 | 9 | 11 | 9
  Temperature: Mild | 0 | 0 | 0 | 0 | 0 | 1
  Temperature: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Any Systemic Symptom: None | 7 | 9 | 9 | 7 | 7 | 6
  Any Systemic Symptom: Mild | 2 | 2 | 2 | 2 | 3 | 4
  Any Systemic Symptom: Moderate | 1 | 0 | 0 | 0 | 1 | 0
  Any Systemic Symptom: Severe | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Subjects Reporting Systemic Reactogenicity Signs and Symptoms Within 7 Days of Any Product Administration of DS-Cav1 Alone or With Alum Adjuvant
Description: Subjects recorded the occurrence of solicited symptoms on a diary card for 7 days after each study product administration and reviewed the diary card with clinic staff at a follow up visit. Subjects were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of subjects reporting any systemic symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA Guidance - September 2007).
Time Frame: 7 days after each product administration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DS-Cav1 (50 mcg) | Group 2: DS-Cav1 (50 mcg) + Alum | Group 3: DS-Cav1 (150 mcg) | Group 4: DS-Cav1 (150 mcg) + Alum | Group 5: DS-Cav1 (500 mcg) | Group 6: DS-Cav1 (500 mcg) + Alum | All DS-Cav1 Dose Groups
Number analyzed (Participants) | 15 | 15 | 20 | 15 | 15 | 15 | 95
Participants
  Malaise: None | 12 | 11 | 17 | 12 | 9 | 11 | 72
  Malaise: Mild | 2 | 4 | 3 | 3 | 6 | 4 | 22
  Malaise: Moderate | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Malaise: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 14 | 12 | 17 | 9 | 12 | 12 | 76
  Myalgia: Mild | 1 | 3 | 3 | 6 | 3 | 3 | 19
  Myalgia: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 12 | 10 | 17 | 9 | 11 | 10 | 69
  Headache: Mild | 3 | 5 | 3 | 6 | 3 | 5 | 25
  Headache: Moderate | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Headache: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 14 | 15 | 20 | 14 | 13 | 13 | 89
  Chills: Mild | 1 | 0 | 0 | 1 | 2 | 2 | 6
  Chills: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 14 | 14 | 19 | 15 | 14 | 13 | 89
  Nausea: Mild | 1 | 1 | 1 | 0 | 1 | 2 | 6
  Nausea: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: None | 15 | 15 | 20 | 15 | 14 | 14 | 93
  Temperature: Mild | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Temperature: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Systemic Symptom: None | 10 | 10 | 13 | 8 | 8 | 7 | 56
  Any Systemic Symptom: Mild | 4 | 5 | 7 | 7 | 6 | 8 | 37
  Any Systemic Symptom: Moderate | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Any Systemic Symptom: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Subjects With Abnormal Laboratory Measures of Safety
Description: Any abnormal laboratory results recorded as unsolicited AEs are summarized. Safety laboratory parameters included hematology (hemoglobin, hematocrit, mean corpuscular volume (MCV), platelets, white blood cell (WBC) and red blood cell (RBC) counts, and neutrophil, lymphocyte, monocyte, eosinophil and basophil percents and counts) and chemistry (alanine aminotransferase (ALT) and creatinine). Complete blood count (CBC) differential, platelet, creatinine and ALT results were collected at screening (≤ 56 days before enrollment), Day 0 prior to study product administration (baseline), and at Days 7, 28, 84, 91 and 112. Institutional laboratory normals as well as the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventative Vaccine Clinical Trials FDA Guidance, September 2007 were used.
Time Frame: Day 0 through Day 308
Population: Population included all enrolled subjects who had laboratory results available at any study visit post baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DS-Cav1 (50 mcg) | Group 2: DS-Cav1 (50 mcg) + Alum | Group 3: DS-Cav1 (150 mcg) | Group 4: DS-Cav1 (150 mcg) + Alum | Group 5: DS-Cav1 (500 mcg) | Group 6: DS-Cav1 (500 mcg) + Alum | All DS-Cav1 Dose Groups
Number analyzed (Participants) | 15 | 15 | 20 | 15 | 15 | 15 | 95
Participants
  ALT | 0 | 1 | 1 | 1 | 0 | 0 | 3
  Creatinine | 0 | 1 | 0 | 0 | 0 | 0 | 1
  WBC Count | 1 | 0 | 0 | 1 | 1 | 0 | 3
  Hemoglobin | 3 | 0 | 1 | 1 | 4 | 1 | 10
  Neutrophil Count | 0 | 2 | 1 | 0 | 2 | 1 | 6
  Lymphocyte Count | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Eosinophil Count | 0 | 0 | 0 | 0 | 1 | 0 | 1

8. Primary Outcome: Number of Subjects With One or More Unsolicited Non-Serious Adverse Events (AEs)
Description: Unsolicited AEs and attribution assessments were recorded in the study database from receipt of the first study product administration through the visit scheduled for 28 days after each study product administration. At other time periods between study product administrations and when greater than 28 days after the last study product administration, only serious AEs (SAEs reported as a separate outcome and in the AE module) and new chronic medical conditions that required ongoing medical management were recorded through the last study visit. The relationship between an AE and the study product was assessed by the investigator on the basis of his or her clinical judgment and the definitions outlined in the protocol. A subject with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through Day 28 after product administration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DS-Cav1 (50 mcg) | Group 2: DS-Cav1 (50 mcg) + Alum | Group 3: DS-Cav1 (150 mcg) | Group 4: DS-Cav1 (150 mcg) + Alum | Group 5: DS-Cav1 (500 mcg) | Group 6: DS-Cav1 (500 mcg) + Alum
Number analyzed (Participants) | 15 | 15 | 20 | 15 | 15 | 15
Participants
  Related to Study Product | 3 | 3 | 2 | 0 | 4 | 3
  Unrelated to Study Product | 3 | 7 | 12 | 7 | 7 | 6

9. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs were reported from receipt of first study product administration through the last expected study visit at Day 308. The relationship between a SAE and the study product was assessed by the investigator on the basis of his or her clinical judgment and the definitions outlined in the protocol. A subject with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through Day 308
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DS-Cav1 (50 mcg) | Group 2: DS-Cav1 (50 mcg) + Alum | Group 3: DS-Cav1 (150 mcg) | Group 4: DS-Cav1 (150 mcg) + Alum | Group 5: DS-Cav1 (500 mcg) | Group 6: DS-Cav1 (500 mcg) + Alum
Number analyzed (Participants) | 15 | 15 | 20 | 15 | 15 | 15
Participants
  Related to Study Product | 0 | 0 | 0 | 0 | 0 | 0
  Unrelated to Study Product | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Subjects Who Had Respiratory Syncytial Virus (RSV) Infection Following Product Administration
Description: Respiratory Syncytial Virus (RSV) cases were recorded in the study database from receipt of the first study product administration through the last study visit.
Time Frame: Day 0 through Day 308
Population: Population included all enrolled subjects who received at least one study injection of DS-Cav1 alone or with alum adjuvant (N=95).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: DS-Cav1 (50 mcg) | Group 2: DS-Cav1 (50 mcg) + Alum | Group 3: DS-Cav1 (150 mcg) | Group 4: DS-Cav1 (150 mcg) + Alum | Group 5: DS-Cav1 (500 mcg) | Group 6: DS-Cav1 (500 mcg) + Alum
Number analyzed (Participants) | 15 | 15 | 20 | 15 | 15 | 15
Participants | 1 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Respiratory Syncytial Virus Subtype A (RSV A) Antigen-specific Neutralizing Antibody Geometric Mean Titers (GMTs) at 4 Weeks After the First Product Administration of DS-Cav1 Alone or With Alum Adjuvant
Description: Neutralizing antibody titers were determined against a reporter RSV A2 virus (RSV A), and were summarized using geometric mean 50% inhibitory concentration (IC50). Negative samples were reported and IC50 titers were calculated using half the limit of detection. Measurements were normalized to international units per milliliter.
Time Frame: 4 weeks after the first product administration (Week 4)
Population: as for outcome 10
Measure: Geometric Mean (Full Range); unit: titer
Arm/Group | Group 1: DS-Cav1 (50 mcg) | Group 2: DS-Cav1 (50 mcg) + Alum | Group 3: DS-Cav1 (150 mcg) | Group 4: DS-Cav1 (150 mcg) + Alum | Group 5: DS-Cav1 (500 mcg) | Group 6: DS-Cav1 (500 mcg) + Alum
Number analyzed (Participants) | 15 | 15 | 20 | 15 | 15 | 15
titer
  Week 0 (Baseline, Pre-Administration) | 777 [192 to 3167] | 689 [288 to 2141] | 736 [216 to 4676] | 653 [186 to 2476] | 707 [230 to 5725] | 669 [321 to 1840]
  Week 4 | 4203 [1001 to 10910] | 3486 [1385 to 18852] | 5422 [2050 to 13104] | 5513 [1715 to 17602] | 7495 [2370 to 16870] | 6083 [2301 to 13522]

12. Secondary Outcome: Respiratory Syncytial Virus Subtype A (RSV A) Antigen-specific Neutralizing Antibody Geometric Mean Titers (GMTs) at 4 Weeks After the Second Product Administration of DS-Cav1 Alone or With Alum Adjuvant
Description: as for outcome 11
Time Frame: 4 weeks after the second product administration (Week 16)
Population: Population included all enrolled subjects who received the optional second study injection of DS-Cav1 alone or with alum adjuvant (N=62).
Measure: Geometric Mean (Full Range); unit: titer
Arm/Group | Group 1: DS-Cav1 (50 mcg) | Group 2: DS-Cav1 (50 mcg) + Alum | Group 3: DS-Cav1 (150 mcg) | Group 4: DS-Cav1 (150 mcg) + Alum | Group 5: DS-Cav1 (500 mcg) | Group 6: DS-Cav1 (500 mcg) + Alum
Number analyzed (Participants) | 10 | 11 | 11 | 9 | 11 | 10
titer
  Week 0 (Baseline, Pre-Administration) | 866 [192 to 3167] | 734 [288 to 2141] | 790 [498 to 1601] | 578 [186 to 1526] | 680 [267 to 1300] | 839 [486 to 1840]
  Week 16 | 3844 [1108 to 9545] | 2536 [1566 to 10771] | 4201 [1985 to 9673] | 4033 [2235 to 7977] | 5193 [2783 to 9251] | 4440 [1909 to 10551]

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs) were reported for 7 days after each study injection. Unsolicited AEs were recorded from receipt of the first study injection through the visit scheduled 4 weeks after each study injection. At other time periods between injections and when greater than 4 weeks after the last injection, only serious AEs and new chronic medical conditions that required ongoing medical management were recorded through the last study visit.
Description: Solicited AEs collected through systematic assessment and unsolicited AEs collected through non-systematic assessment are reported by subjects who received at least one study injection and provided safety data following the injection, and represent the number and percentage of subjects reporting the event. A subject with multiple experiences of the same event is counted once using the event of worst severity.
Arm/Group | Group 1: DS-Cav1 (50 mcg) | Group 2: DS-Cav1 (50 mcg) + Alum | Group 3: DS-Cav1 (150 mcg) | Group 4: DS-Cav1 (150 mcg) + Alum | Group 5: DS-Cav1 (500 mcg) | Group 6: DS-Cav1 (500 mcg) + Alum
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/20 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/20 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 12/15 | 12/15 | 20/20 | 13/15 | 14/15 | 12/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: DS-Cav1 (50 mcg) (N=15) | Group 2: DS-Cav1 (50 mcg) + Alum (N=15) | Group 3: DS-Cav1 (150 mcg) (N=20) | Group 4: DS-Cav1 (150 mcg) + Alum (N=15) | Group 5: DS-Cav1 (500 mcg) (N=15) | Group 6: DS-Cav1 (500 mcg) + Alum (N=15)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 1 | 1 | 4 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 2 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 4 | 7 | 2 | 2 | 3
Administration site pain (General disorders) | 11 | 10 | 12 | 12 | 11 | 12
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Burns first degree (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 5 | 3 | 6 | 4 | 5
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1 | 2
Administration site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 1 | 0 | 0 | 1 | 2 | 2
Malaise (General disorders) | 3 | 4 | 3 | 3 | 6 | 4
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 6 | 3 | 3
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/88/NCT03049488/Prot_SAP_ICF_000.pdf